CLINICAL TRIAL: NCT02086409
Title: Dairy Product, Calcium & Vitamin D Supplementation and Cognitive-motor Function
Brief Title: GAit, MEmory, Dietary and Vitamin D
Acronym: GAME-D2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-A01499-36
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2014-03

CONDITIONS: Memory Complaint Without Cognitive Decline
MeSH Terms: interventions — Vitamin D; Calcium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yogurt supplemented with vitamin D and calcium (Experimental): 20 participants take yogurt supplemented with vitamin D and calcium during 12 weeks
  Interventions: Dietary Supplement: Yogurt supplemented with vitamin D and calcium
- Yogurt not supplemented with vitamin D and calcium (Active Comparator): 20 participants take yogurt not supplemented with vitamin D and calcium during 12 weeks
  Interventions: Dietary Supplement: Yogurt not supplemented with vitamin D and calcium

INTERVENTIONS:
Dietary Supplement: Yogurt supplemented with vitamin D and calcium — The product is a yogurt containing 200 IU of vitamin D and 400 mg of calcium. Participants take 2 yogurts per day.
  Arms: Yogurt supplemented with vitamin D and calcium
Dietary Supplement: Yogurt not supplemented with vitamin D and calcium — The comparator is represented by a yogurt not supplemented with vitamin D and calcium.Participants take 2 yogurts per day.
  Arms: Yogurt not supplemented with vitamin D and calcium

SUMMARY:
Gait and posture disorders are very common in subjects aged 65 and over, and result mainly from neuromuscular and cognitive disorders.

Many studies have shown that 1) vitamin D deficiency is very common in women aged 65 and over, 2) individuals with hypovitaminosis D have lower muscle, gait and executive performances and are more prone to fail than individuals with no hypovitaminosis D, 3) the intake of vitamin D combined or not with calcium may improve muscle strength and cognitive performance.

The investigators hypothesized that the daily intake of 2 yogurts containing 200 IU of vitamin D and 400 mg of calcium 1) can improve spatiotemporal gait parameters, posture and executive performance, 2) and that this improvement depends of the initial level of vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 65 and over
* To have hypovitaminosis D (i.e. serum 25-hydroxyvitamin D [25OHD] concentration ≤ 30ng/mL)
* To have no hypercalcemia (defined as serum calcium concentration ≥ 2,65mmol/L)
* Ability to walk a distance of 15 meters unaided
* Ability to eat 2 yogurts per day
* Memory complaint without cognitive decline
* To have given and signed an informed consent to participate in the trial
* To be affiliated to French Social Security
* To have no vitamin D supplementation during inclusion

Exclusion Criteria:

* Existence of dementia according to DSM-IV and NINCDS-ADRDA criteria and others cognitive disorders: untreated thyroid dysfunction, chronic ongoing ethylism, history of syphilis, stroke with sequelae, depressive symptomatology (Geriatric Depression Scale > 5/15)
* Osteoarticular diseases of the lower members and / or spine altering the biomechanical characteristics of the body.
* Vitamin D supplementation during inclusion
* Contraindications to vitamin D
* Unstable medical condition
* Dairy allergy
* Taste of dairy products not supported
* Enrolment in another simultaneous clinical trial
* Civil defense measures underway
* Refusal to participate of the subject

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in spatiotemporal gait, and in particular in the variability of stride time | This outcome is assessed at baseline and 12 weeks after oral intake.
  Stride time variability is measured with spatiotemporal analysis of walking

SECONDARY OUTCOMES:
Change in posture | This outcome is assessed at baseline and 12 weeks after oral intake.
  Posture is evaluated with Time Up & Go, Five Time Sit-to-Stand and posture analysis with a platform.
Change in grip strength | This outcome is assessed at baseline and 12 weeks after oral intake.
  Grip strength is measured with a dynamometer.
Change in executive performance | This outcome is assessed at baseline and 12 weeks after oral intake.
  Executive performance is measured with Trial Making Test part B (TMT B)
Change in other cognitive scores | These outcomes are assessed at baseline and 12 weeks after oral intake.
  Executive scores are assessed with digit span test (forward and backward), Trial Making Test part A (TMT A), Stoop test and Processing Speed Index
Change in the serum concentration of 25 OHD | This outcome is assessed at baseline and 12 weeks after oral intake.
  This outcome is assessed with the serum concentrations of 25OHD
Compliance to intervention | This outcome is assessed 12 weeks after oral intake.
  Compliance is measured by the number of yogurt capsules returned

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Angers, Angers, Maine et Loire, France